CLINICAL TRIAL: NCT06326346
Title: A Phase II Study of Oral Paclitaxel (Liporaxel) in GIST Patients With a Low P-glycoprotein Expression After Failure With Imatinib, Sunitinib and Regorafenib
Brief Title: GIST Oral Paclitaxel(Liporaxel)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2401
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Paclitaxel (Liporaxel) (Experimental): Liporaxel 200mg/m2 twice daily orally on day 1, 8, and 15 every 4 weeks (1 cycle = 4 weeks)
  Interventions: Drug: Liporaxel

INTERVENTIONS:
Drug: Liporaxel — Liporaxel 200mg/m2 twice daily orally on day 1, 8, and 15 every 4 weeks (1 cycle = 4 weeks)

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Liporaxel for patients with GIST who failed on prior standard treatments, including imatinib, sunitinib, and regorafenib, and with low P-glycoprotein expression.

DETAILED DESCRIPTION:
The survival outcomes of patients with advanced and/or metastatic gastrointestinal stromal tumors (GIST) have markedly improved with application of imatinib, the KIT tyrosine kinase inhibitor (GlivecTM, Novartis) for the treatment. Recently, sunitinib (SuteneTM, Pfizer) and regorafenib (StivargaTM, Bayer) have shown efficacy in patients with disease progression on imatinib as second- and third-line treatment, respectively. However, most patients develop acquired resistance to KIT tyrosine kinase inhibitors and show disease progression.

While cytotoxic chemotherapeutic agents were expected to have minimal antitumor effect on GIST, recent preclinical studies have shown that 37 out of 89 different chemotherapeutic agents have shown antitumor effects on at least one or more GIST cell lines. Especially, topoisomerase II inhibitors, paclitaxel, bortezomib have shown promising results. Based on the results, the investigators conducted a single center, single arm phase II study to evaluate efficacy and safety of paclitaxel for patients with GIST who failed to prior imatinib and sunitinib. Overall efficacy was modest, although patients with low P-glycoprotein expression showed better efficacy compared to those with high P-glycoprotein expression. Subsequently, the investigators performed another phase 2 trial to evaluate efficacy of paclitaxel for previously treated GIST patients with low P-glycoprotein expression and have met the primary endpoint.

Liporaxel is an oral formulation of paclitaxel, and showed high bioavailability, safety, and antitumor effect from non-clinical studies. From a phase 1 clinical trial for metastatic solid tumor patients, Liporaxel showed adequate PK/PD profiles. Compared to intravenous paclitaxel, administration is relatively easier and has better safety in terms of hypersensitivity reaction which is caused by the admixture of intravenous formulation of paclitaxel. From a multicenter phase 3 trial conducted in South Korea for patients with advanced gastric adenocarcinoma who failed on first-line palliative chemotherapy (DREAM trial), Liporaxel showed non-inferiority compared to intravenous paclitaxel in terms of both safety and efficacy, and it is currently approved for the second-line treatment in advanced gastric cancer. Also, Liporaxel proved safety and potential efficacy in patients with HER2 negative metastatic breast cancer as first-line chemotherapy, and currently multicenter phase 3 trial in ongoing (OPTIMAL3 trial).

The purpose of this study is to evaluate safety and efficacy of Liporaxel for patients with GIST who failed on prior standard treatments, including imatinib, sunitinib, and regorafenib, and with low P-glycoprotein expression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or older, at the time of acquisition of informed consent
2. Histologically confirmed metastatic and/or advanced GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
3. Failed (progressed and/or intolerable) after prior treatments for GIST, including at least imatinib and sunitinib, regorafenib.
4. Adequate tissue obtained after treatment failure to imatinib, sunitinib, and regorafenib for P-glycoprotein immunohistochemistry (IHC) analysis, and showed P-glycoprotein expression of less than 6. (For patients with PDGFRα D842V mutation or other subtypes with poor response to tyrosine kinase inhibitors, tumor tissue obtained at any period can be used.)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0~2
6. Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-CTCAE version 5.0
7. At least one measurable lesion as defined by RECIST version 1.1.
8. Adequate bone marrow, hepatic, renal, and other organ functions

   * Neutrophil >1,500/mm3
   * Platelet > 100,000/mm3
   * Hemoglobin >8.0 g/dL
   * Total bilirubin < 1.5 x upper limit of normal (ULN)
   * AST/ALT < 2.5 x ULN
   * Creatinine <1.5 x ULN
9. Life expectancy > 12 weeks
10. Washout period of previous TKIs or chemotherapy for more than 4 times the half life ((Imatinib and regorafenib need 1 week and sunitinib need 2 weeks.)
11. Provision of a signed written informed consent

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breast feeding
2. Women or men who are not willing to use effective contraception entering the study period or until at least 3 months after the last study drug administration.
3. If any of the following applies within ≤ 6 months prior to starting study enrollment : Myocardial Infarction, severe instable angina, coronary/peripheral bypass, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, treatment required severe arrhythmia.
4. Uncontrolled infection
5. Diabetes mellitus with clinically significant peripheral artery disease
6. Acute and chronic liver disease and all chronic liver impairment.(But Patients with stable chronic hepatitis B are eligible)
7. Uncontrolled gastrointestinal toxicities with toxicity greater than NCI CTCAE grade 2
8. Acute, or chronic medical or psychiatric condition or laboratory abnormality such as active uncontrolled infection that difficult to study participation in the judgment of the investigator
9. The patient experienced any bleeding episode considered life-threatening, or any grade 3 or 4 bleeding event. (required transfusion or endoscopic or surgical intervention)
10. Patient who underwent major surgery or is under recovery from surgery within 28 days from the study treatment
11. Known diagnosis of HIV infection (HIV testing is not mandatory).
12. History of another primary malignancy that is currently clinically significant or currently requires active intervention.
13. Patients with clinically suspected brain metastasis symptom, brain metastases as assessed by radiologic imaging.
14. Alcohol or substance abuse disorder.
15. Known severe hypersensitivity to paclitaxel
16. Received paclitaxel-based treatment for GIST

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
16 week disease control rate | 16 weeks
  according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Progression-free survival | until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  time from the date of first administration of palliative first-line chemotherapy to the date of the first objectively documented tumor progression or death, whichever occurs first)
Overall survival | through study completion, an average of 3 years
  time from the date of first administration of palliative first-line chemotherapy to the date of death due to any cause
Objective response rate | every 4 weeks for the initial two evaluation, then every 8 weeks
  according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Adverse event assessed by NCI-CTCAE Version 5.0 | until 28 days from the last administration of the investigational product
  assessed by NCI-CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpagu, South Korea

IPD SHARING:
Plan to Share IPD: No